CLINICAL TRIAL: NCT03172299
Title: Prevention of Neovascular Glaucoma by Intravitreal Injections of Anti-Vascular Endothelial Growth Factor in Patients Treated with Proton Therapy for a Large Choroidal Melanoma
Brief Title: Prevention of Neovascular Glaucoma by Intravitreal Injections of Anti-VEGF in Patients Treated with Proton Therapy for a Large Choroidal Melanoma
Acronym: PROTECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-API-01
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Ocular Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Injection of anti-VEGF (Active Comparator)
  Interventions: Drug: Aflibercept Injection
- false injection of anti-VEGF (Placebo Comparator)
  Interventions: Drug: False injection

INTERVENTIONS:
Drug: Aflibercept Injection — Intravitreal injection of aflibercept 40mg/mL will be done on patients. The injections will be performed on the last day of the proton therapy, then 1 and 2 months later for the induction phase. During the maintenance phase, injections will be performed every 3 months for a period of 21 months.
  Arms: Injection of anti-VEGF
Drug: False injection — A false injection will be done on patients on the last day of the proton therapy, then 1 and 2 months later for the induction phase. During the maintenance phase, falses injections will be performed every 3 months for a period of 21 months.
  Arms: false injection of anti-VEGF

SUMMARY:
The reference treatment of ocular melanoma is a conservative treatment by proton therapy. Its goal is to treat the tumor while preserving the eyeball and visual acuity. However, ablation of the eyeball is sometimes necessary after proton therapy in the case of neovascular glaucoma. This complication occurs in 7 to 47% of cases (depending on the size of the tumor) and is associated with hypersecretion of Vascular Endothelial Growth Factor (VEGF) related to necrotic and inflammatory tumor tissue after proton therapy or ischemic retina. The intravitreal injections of anti-VEGF are used in the treatment of neovascular radicular glaucoma without avoiding enucleation in all cases. The investigators propose to study the prevention of neovascular glaucoma by intravitreal prophylactic administration of anti-VEGF.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Choroid melanoma more than 7mm thick and / or over basal diameter of 15mm treated by proton therapy

Exclusion Criteria:

* Iris melanoma
* Melanoma immediately metastatic
* Pregnant or breastfeeding women
* Known hypersensitivity to aflibercept (anti-VEGF selected)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of neovascular glaucoma | at 5 years
  Occurrence of neovascular glaucoma after radiation-induced proton therapy. Clinical diagnosis (examination at the slit lamp)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie BAILLIF, Pr, Study Director — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No